CLINICAL TRIAL: NCT02818855
Title: Treatment of Multiple Gingival Recessions With Collagen Matrix Versus Subepithelial Connective Tissue Graft: A Non-inferiority Randomized Clinical Trial
Brief Title: Treatment of Multiple Gingival Recessions
Acronym: 3DMUCO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Chairperson, Department of Periodontics, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3DMUCO
Record Dates: First submitted 2013-08-20; First posted 2016-06-30 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Gingival Recession
Keywords: Root coverage; Gingival recession; Plastic surgery; Connective tissue graft; Mucograft
MeSH Terms: conditions — Gingival Recession | interventions — Mucograft

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collagen Matrix plus coronally advanced flap (CAF) (Experimental): A new collagen matrix (Mucograft) associated to coronally advanced flap
  Interventions: Procedure: Coronally advanced flap (CAF); Drug: Collagen Matrix
- Subepithelial connective tissue graft plus CAF (Active Comparator): Subepithelial connective tissue graft associated to coronally advanced flap
  Interventions: Procedure: Coronally advanced flap (CAF); Procedure: Subepithelial connective tissue graft

INTERVENTIONS:
Procedure: Coronally advanced flap (CAF) — The test group will be treated by means of the association of Collagen Matrix + Coronally Advanced Flap. As treatment, the control group will receive the association of a subepithelial Conjunctive Tissue Graft + Coronally Advanced Flap.
  The aim of both procedures will be to obtain root coverage. All these procedures will be performed in a standardized manner.
  Other Names: Subepithelial conjunctive tissue grafts; Coronally advanced flaps; Coronally advanced flaps associated with collagen matrix
Drug: Collagen Matrix — A new collagen membrane
  Other Names: Mucograft
  Arms: Collagen Matrix plus coronally advanced flap (CAF)
Procedure: Subepithelial connective tissue graft — Connective tissue graft
  Other Names: connective tissue graft
  Arms: Subepithelial connective tissue graft plus CAF

SUMMARY:
Gingival recession (GR) is frequently associated with deterioration in dental esthetics and dental hypersensitivity. Outcomes from recent systematic reviews have demonstrated that when the root is covered and the gain in the width of keratinized tissue (KT) is expected, the use of subepithelial connective tissue grafts (SCTGs) associated with coronally advanced flaps (CAF) appears to be more predictable, and may be considered the gold standard procedure. However, the SCTGs may increase patients' morbidity (e.g., pain). This occurs because of the need for a donor surgical area, which may increase the risk of surgical complications like bleeding, as well as increases post-operative discomfort and the period of the surgical procedure. Another biomaterial, a new collagen matrix (CM) has been used as a substitute for the SCTG. The use of CM was associated with a significant reduction in post-operative morbidity, less post-operative pain and discomfort in the patient, and more esthetic satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be included in the study if they fulfill the following inclusion criteria:

  1. a clinical diagnosis of multiple-recession type defects at maxillary canines and premolars with at least one GR ≥ 3mm in depth;
  2. areas of Miller's Class I or II GR;
  3. teeth without root abrasions or caries.

Exclusion Criteria: -

The exclusion criteria used will be as follows:

* patients allergic to collagen
* a history of smoking (within the previous 6 months)
* pregnancy or lactation
* a history of destructive periodontal disease or the formation of recurrent abscesses
* root caries at the site of recession
* previous surgical root coverage procedures
* systemic healing disorders (for example, acquired immunodeficiency syndrome [AIDS], diabetes mellitus or risk factors evaluated by a medical doctor)
* periodontal disease, or poor plaque control (full mouth plaque index > 20%).

The exclusion criteria for teeth will be:

1. noncarious cervical lesions (erosion, abfraction etc.)
2. any type of previous cervical restoration
3. extrusion
4. giroversion
5. mobility
6. a prominent root surface.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage (RC) | 12-months
  The primary clinical outcome will be percentage of root coverage (RC) at 12 months

SECONDARY OUTCOMES:
Reductions in recession depth (RRD) | At the baseline, 3-month, 6-month and 12-months
  Measured from the cementum-enamel junction (CEJ) up to the highest point of the gingival margin
Complete root coverage of the gingival recessions (CRC) | At the baseline, 3-month, 6-month and 12-months
Recession width (RW) at the cemento-enamel junction | At the baseline, 3-month, 6-month and 12-months
Relative clinical attachment level (RCAL) | At the baseline, 3-month, 6-month and 12-months
  Measured from a fixed point (stent) prepared on the acrylic guide up to the base of the gingival sulcus.
Probing depth (PD) | At the baseline, 3-month, 6-month and 12-months
  Calculated as RCAL- PD;
keratinized tissue width (KT) | At the baseline, 3-month, 6-month and 12-months
  From the free gingival margin to the mucogingival junction.
Gain in thickness of gingival tissue (GT) | At the baseline, 3-month, 6-month and 12-months
  With an injection needle and a silicon marker, 2mm below the gingival margin.

OTHER OUTCOMES:
Subject esthetic satisfaction by participants | 1, 3, 6 months and after 12 months
  The participants will be invited to reply to a questionnaire on subject esthetic satisfaction with the surgical results (from dissatisfied to very satisfied) on a scale of 1-5, as well as after 1, 3, 6 months and after 12 months.
Subjective symptoms of pain and discomfort by participants | At 1, 2, 3-week, 1 month, 3-month, 6-month and12-months.
  Subjective symptoms of pain and discomfort (without pain and with a great deal of pain) will be evaluated with 10 cm (0-10) visual analog scales (VAS) at 1, 2, 3-week, 1 month, 3-month, 6-month and12-months.
Esthetic questionnaire by experienced periodontist | 1, 2, 3-week, 1-month, 3-month, 6-month and 12-months after surgery
  One experienced periodontist will be invited to observe the initial photographs and those of the clinical results obtained during the entire healing process and asked to respond to an esthetic questionnaire (from dissatisfied to very satisfied) on a scale of 1 to 5 points after 1, 2, 3-week, 1-month, 3-month, 6-month and 12-months.12 All this examinations also will be performed in the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Romito, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Jepsen K, Jepsen S, Zucchelli G, Stefanini M, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M. Treatment of gingival recession defects with a coronally advanced flap and a xenogeneic collagen matrix: a multicenter randomized clinical trial. J Clin Periodontol. 2013 Jan;40(1):82-9. doi: 10.1111/jcpe.12019. Epub 2012 Oct 10. PMID 23050490
- [Result] McGuire MK, Scheyer ET. Xenogeneic collagen matrix with coronally advanced flap compared to connective tissue with coronally advanced flap for the treatment of dehiscence-type recession defects. J Periodontol. 2010 Aug;81(8):1108-17. doi: 10.1902/jop.2010.090698. PMID 20350159
- [Result] Sanz M, Lorenzo R, Aranda JJ, Martin C, Orsini M. Clinical evaluation of a new collagen matrix (Mucograft prototype) to enhance the width of keratinized tissue in patients with fixed prosthetic restorations: a randomized prospective clinical trial. J Clin Periodontol. 2009 Oct;36(10):868-76. doi: 10.1111/j.1600-051X.2009.01460.x. Epub 2009 Aug 12. PMID 19678861